CLINICAL TRIAL: NCT01610986
Title: Effects of Glucose-fructose Drinks During Training on Lactate Transport and Oxidation and on Endurance Performance
Brief Title: Effects of Glucose-fructose Drinks During Training on Lactate Transport
Acronym: LactEx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Luc Tappy, MD, Professor of Physiology, University of Lausanne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 251/11
Record Dates: First submitted 2012-05-23; First posted 2012-06-04 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Normal Physiology on Healthy Subjects
Keywords: Fructose; Exercise; Lactic acid; Monocarboxylic Acid Transporters
MeSH Terms: conditions — Motor Activity | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose-fructose (Experimental): Participants will take glucose-fructose drinks during training sessions
  Interventions: Dietary Supplement: Glucose-fructose
- Water (Experimental): Participants will take only water during training sessions
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Glucose-fructose — 0.8 g/h glucose and 0.5 g/h fructose during training
  Arms: Glucose-fructose
Dietary Supplement: Water — Only water intake during training
  Arms: Water

SUMMARY:
The purpose of this study is to determine whether glucose-fructose intake during training increases lactate transport and oxidation and improve endurance performance.

DETAILED DESCRIPTION:
The study will enroll 24 healthy male volunteers. After baseline assessment of lactate transport and endurance performance, subjects will be randomized to either a 3-week intervention arm in which they will train with glucose-fructose intake during training, or to a control arm (water during training). After this 3-week intervention, lactate transport and endurance performance will be assessed again.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* age between 18 and 30 years
* sedentary
* BMI between 19 and 25
* blood pressure lower than 140/90 mmHg

Exclusion Criteria:

* smoking
* consumption of more than 10g alcohol per day
* cardiovascular history
* electrographic abnormalities at rest
* consumption of more than one can of soda per day or more than 60g sugars per day
* any current drug treatment
* consumption of drugs or illicit substances
* diabetes mellitus
* vegetarian
* food intolerance
* blood donation or participation to another study <3 months before study inclusion

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in lactate transport | At baseline (before training) and after the 3-week training protocol
  Measurement of lactate production, utilization, oxidation and clearance during a 90 min cycling exercise at 50% VO2 max (measured with 13C-lactate)

SECONDARY OUTCOMES:
Change in muscle monocarboxylate transporters (MCTs) expression and protein content | At baseline (before training) and after the 3-week training protocol
  MCTs expression (mRNA) and protein content after muscle biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Luc Tappy, Pr, Principal Investigator — University of Lausanne
Locations (1):
- University of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Background] Lecoultre V, Benoit R, Carrel G, Schutz Y, Millet GP, Tappy L, Schneiter P. Fructose and glucose co-ingestion during prolonged exercise increases lactate and glucose fluxes and oxidation compared with an equimolar intake of glucose. Am J Clin Nutr. 2010 Nov;92(5):1071-9. doi: 10.3945/ajcn.2010.29566. Epub 2010 Sep 8. PMID 20826630